CLINICAL TRIAL: NCT05291299
Title: Anti-Inflammatory Dietary Intervention for Rheumatoid Arthritis
Acronym: RA-Diet
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Attune Health Research, Inc. (Industry)
Collaborators: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Swamy Venuturupalli, Principal Investigator, Attune Health Research, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 227188
Record Dates: First submitted 2022-01-27; First posted 2022-03-22 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (Control Group) (Other): Physicians will follow standard of care and instruct participants in the control group to follow a Mediterranean diet higher in vegetables and fruits[19]. Patients will be provided with a handout detailing the basics of the Mediterranean diet. At follow up visits, physicians will ask participants about how they have been eating and if they have been following the guidelines.
  Interventions: Other: Control/Standard of Care
- Anti-inflammatory Diet (Intervention Group) (Experimental): An 8-week nutrition program consisting of an individualized elimination diet and systematic food reintroduction implemented and supervised by a Registered Dietitian. Clinical trials have shown some benefit from elimination diets for individuals with autoimmune disease [18].
  The specifics of the elimination diet including duration and foods included will be individual and up to the RDs discretion based on the patient's medical and diet history, willingness, current diet, preferences, goals, and ability. The initial diet instruction with a Registered Dietitian will be a one-hour, individual secure video call, with nutrition evaluation/assessment and education on elimination diet protocol. Follow up visits will be approximately 20-30 minutes for the subsequent 7 weeks.
  Interventions: Behavioral: Anti-inflammatory diet

INTERVENTIONS:
Behavioral: Anti-inflammatory diet — Patients randomized to the intervention group will work with a registered dietitian to create an individualized diet program to help reduce inflammation and Rheumatoid arthritis related symptoms.
  Arms: Anti-inflammatory Diet (Intervention Group)
Other: Control/Standard of Care — Patients randomized to the control group will be following standard of care where their doctor will instruct them to follow a Mediterranean diet and provides them with an instructional sheet.
  Arms: Standard of Care (Control Group)

SUMMARY:
The primary objective of this study is to assess if there is a significant difference in the mean disease activity score in individuals with RA participating in a dietary intervention compared to those in the control group measured by DAS-28. Other measures to track disease activity will include monitoring number and severity of disease flares and any changes in medications. This will be done by completing a single-blinded randomized controlled trial, parallel in design. The study population will consist of adults diagnosed with Seropositive and Seronegative RA based on the American College of Rheumatology criteria. Participants will have low, moderate, or high disease activity based on DAS-28 where the investigator feels that they can see improvement from a dietary intervention.

DETAILED DESCRIPTION:
Per the Schedule of Assessments, upon enrollment, participants will be required to come in for a total of five on site visits. The first visit, also known as the baseline visit, will require participants to provided informed consent after all eligibility criteria is met. Subsequently, participants' Demographics, Medical History, EULAR/ACR classification, and physicians' assessments will be documented. Participants' vital signs will be checked and a thorough physical exam will also be performed after which safety labs will be drawn in addition to a routine urinalysis. Participants will complete outcome surveys and a food frequency questionnaire. Participants' body composition will be measured. Concomitant medications will be reviewed. Each participant will receive nutrition education from an approved MD or a consultation with an approved RD depending on the group to which they have been randomized. Participants who receive consultations with an RD will have seven follow up visits after the baseline visit.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years.
* Diagnosed RA by a rheumatologist determined by the 2010 ACR/EULAR Classification Criteria.
* Low, moderate, or highly active disease state based on clinical assessment where the investigator feels there is potential to see a difference.
* Able to read and write in English.

Exclusion Criteria:

* Younger than 18 years.
* Unable to attend the 8 weekly nutrition appointment.
* History of documented eating disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2022-07-05 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Disease Activity | 8 weeks
  Rheumatoid arthritis disease activity Measured by Disease Activity Score-28, higher score is associated with increased disease activity. a Disease Activity Score greater than 5.1 indicated very active disease while a Disease Activity Score that is lower than 2.6 indicates disease remission
Disease Activity | 52 weeks
  Rheumatoid arthritis disease activity Measured by Disease Activity Score-28, higher score is associated with increased disease activity. a Disease Activity Score greater than 5.1 indicated very active disease while a Disease Activity Score that is lower than 2.6 indicates disease remission

SECONDARY OUTCOMES:
Patient reported outcomes | 8 weeks
  change in patient reported disease related outcomes measured by Health Assessment Questionaire-Disability Index, where a higher score indicates lower quality of health. A 0 indicates no difficulty in task performance while a score of 3 indicates much difficulty in task performance
Patient reported outcomes | 52 weeks
  change in patient reported disease related outcomes measured by Health Assessment Questionaire-Disability Index, where a higher score indicates lower quality of health. A 0 indicates no difficulty in task performance while a score of 3 indicates much difficulty in task performance
Patient reported outcomes | 8 weeks
  change in patient reported disease related outcomes measured by Physical and Mental Health Summary Score (PROMIS-29) where a score of 0 indicates excellent mental and physical health while a score of 10 indicates poor mental and physical health.
Patient reported outcomes | 52 weeks
  change in patient reported disease related outcomes measured by Physical and Mental Health Summary Score (PROMIS-29) where a score of 0 indicates excellent mental and physical health while a score of 10 indicates poor mental and physical health.
Anthropometric measurements | 8 weeks
  Assess the change in anthropometric measurements by weight
Anthropometric measurements | 52 weeks
  Assess the change in anthropometric measurements by weight
Anthropometric measurements | 8 weeks
  Assess the change in anthropometric measurements by body fat percentage (waist circumference)
Anthropometric measurements | 52 weeks
  Assess the change in anthropometric measurements by body fat percentage (waist circumference)
Anthropometric measurements | 8 weeks
  Assess the change in anthropometric measurements by waist/hip ratio
Anthropometric measurements | 52 weeks
  Assess the change in anthropometric measurements by waist/hip ratio

CONTACTS AND LOCATIONS:
Locations (1):
- Attune Health Research Inc, Beverly Hills, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chen YM, Chen HH, Hsieh CW, Hsieh TY, Lan JL, Chen DY. A close association of body cell mass loss with disease activity and disability in Chinese patients with rheumatoid arthritis. Clinics (Sao Paulo). 2011;66(7):1217-22. doi: 10.1590/s1807-59322011000700016. PMID 21876977
- [Background] Tajik N, Frech M, Schulz O, Schalter F, Lucas S, Azizov V, Durholz K, Steffen F, Omata Y, Rings A, Bertog M, Rizzo A, Iljazovic A, Basic M, Kleyer A, Culemann S, Kronke G, Luo Y, Uberla K, Gaipl US, Frey B, Strowig T, Sarter K, Bischoff SC, Wirtz S, Canete JD, Ciccia F, Schett G, Zaiss MM. Targeting zonulin and intestinal epithelial barrier function to prevent onset of arthritis. Nat Commun. 2020 Apr 24;11(1):1995. doi: 10.1038/s41467-020-15831-7. PMID 32332732
- [Background] de Carvalho MR, Tebexreni AS, Salles CA, Barros Neto T, Natour J. Oxygen uptake during walking in patients with rheumatoid arthritis--a controlled study. J Rheumatol. 2004 Apr;31(4):655-62. PMID 15088289
- [Background] Guerreiro CS, Calado A, Sousa J, Fonseca JE. Diet, Microbiota, and Gut Permeability-The Unknown Triad in Rheumatoid Arthritis. Front Med (Lausanne). 2018 Dec 14;5:349. doi: 10.3389/fmed.2018.00349. eCollection 2018. PMID 30619860
- [Background] Zhong D, Wu C, Zeng X, Wang Q. The role of gut microbiota in the pathogenesis of rheumatic diseases. Clin Rheumatol. 2018 Jan;37(1):25-34. doi: 10.1007/s10067-017-3821-4. Epub 2017 Sep 15. PMID 28914372
- [Background] Paolino S, Pacini G, Patane M, Alessandri E, Cattelan F, Goegan F, Pizzorni C, Gotelli E, Cutolo M. Interactions between microbiota, diet/nutrients and immune/inflammatory response in rheumatic diseases: focus on rheumatoid arthritis. Reumatologia. 2019;57(3):151-157. doi: 10.5114/reum.2019.86425. Epub 2019 Jun 28. PMID 31462830
- [Background] Gioia C, Lucchino B, Tarsitano MG, Iannuccelli C, Di Franco M. Dietary Habits and Nutrition in Rheumatoid Arthritis: Can Diet Influence Disease Development and Clinical Manifestations? Nutrients. 2020 May 18;12(5):1456. doi: 10.3390/nu12051456. PMID 32443535
- [Background] Leeming ER, Johnson AJ, Spector TD, Le Roy CI. Effect of Diet on the Gut Microbiota: Rethinking Intervention Duration. Nutrients. 2019 Nov 22;11(12):2862. doi: 10.3390/nu11122862. PMID 31766592
- [Background] Camilleri M, Lyle BJ, Madsen KL, Sonnenburg J, Verbeke K, Wu GD. Role for diet in normal gut barrier function: developing guidance within the framework of food-labeling regulations. Am J Physiol Gastrointest Liver Physiol. 2019 Jul 1;317(1):G17-G39. doi: 10.1152/ajpgi.00063.2019. Epub 2019 May 24. PMID 31125257
- [Background] Kjeldsen-Kragh J, Haugen M, Borchgrevink CF, Laerum E, Eek M, Mowinkel P, Hovi K, Forre O. Controlled trial of fasting and one-year vegetarian diet in rheumatoid arthritis. Lancet. 1991 Oct 12;338(8772):899-902. doi: 10.1016/0140-6736(91)91770-u. PMID 1681264
- [Background] Khanna S, Jaiswal KS, Gupta B. Managing Rheumatoid Arthritis with Dietary Interventions. Front Nutr. 2017 Nov 8;4:52. doi: 10.3389/fnut.2017.00052. eCollection 2017. PMID 29167795
- [Background] Aletaha D, Neogi T, Silman AJ, Funovits J, Felson DT, Bingham CO 3rd, Birnbaum NS, Burmester GR, Bykerk VP, Cohen MD, Combe B, Costenbader KH, Dougados M, Emery P, Ferraccioli G, Hazes JM, Hobbs K, Huizinga TW, Kavanaugh A, Kay J, Kvien TK, Laing T, Mease P, Menard HA, Moreland LW, Naden RL, Pincus T, Smolen JS, Stanislawska-Biernat E, Symmons D, Tak PP, Upchurch KS, Vencovsky J, Wolfe F, Hawker G. 2010 Rheumatoid arthritis classification criteria: an American College of Rheumatology/European League Against Rheumatism collaborative initiative. Arthritis Rheum. 2010 Sep;62(9):2569-81. doi: 10.1002/art.27584. PMID 20872595
- [Background] Shadick NA, Sowell NF, Frits ML, Hoffman SM, Hartz SA, Booth FD, Sweezy M, Rogers PR, Dubin RL, Atkinson JC, Friedman AL, Augusto F, Iannaccone CK, Fossel AH, Quinn G, Cui J, Losina E, Schwartz RC. A randomized controlled trial of an internal family systems-based psychotherapeutic intervention on outcomes in rheumatoid arthritis: a proof-of-concept study. J Rheumatol. 2013 Nov;40(11):1831-41. doi: 10.3899/jrheum.121465. Epub 2013 Aug 15. PMID 23950186
- [Background] Darlington LG, Ramsey NW, Mansfield JR. Placebo-controlled, blind study of dietary manipulation therapy in rheumatoid arthritis. Lancet. 1986 Feb 1;1(8475):236-8. doi: 10.1016/s0140-6736(86)90774-9. PMID 2868255
- [Background] Anderson J, Caplan L, Yazdany J, Robbins ML, Neogi T, Michaud K, Saag KG, O'Dell JR, Kazi S. Rheumatoid arthritis disease activity measures: American College of Rheumatology recommendations for use in clinical practice. Arthritis Care Res (Hoboken). 2012 May;64(5):640-7. doi: 10.1002/acr.21649. PMID 22473918
- [Background] Deyo RA, Katrina Ramsey, Buckley DI, Michaels L, Kobus A, Eckstrom E, Forro V, Morris C. Performance of a Patient Reported Outcomes Measurement Information System (PROMIS) Short Form in Older Adults with Chronic Musculoskeletal Pain. Pain Med. 2016 Feb;17(2):314-24. doi: 10.1093/pm/pnv046. PMID 26814279
- [Background] Bigaard J, Frederiksen K, Tjonneland A, Thomsen BL, Overvad K, Heitmann BL, Sorensen TI. Waist circumference and body composition in relation to all-cause mortality in middle-aged men and women. Int J Obes (Lond). 2005 Jul;29(7):778-84. doi: 10.1038/sj.ijo.0802976. PMID 15917857
- [Background] Konijn NP, van Tuyl LH, Bultink IE, Lems WF, Earthman CP, van Bokhorst-de van der Schueren MA. Making the invisible visible: bioelectrical impedance analysis demonstrates unfavourable body composition in rheumatoid arthritis patients in clinical practice. Scand J Rheumatol. 2014;43(4):273-8. doi: 10.3109/03009742.2013.852239. Epub 2014 Feb 7. PMID 24797672
- [Background] Thompson FE, Subar AF, Brown CC, Smith AF, Sharbaugh CO, Jobe JB, Mittl B, Gibson JT, Ziegler RG. Cognitive research enhances accuracy of food frequency questionnaire reports: results of an experimental validation study. J Am Diet Assoc. 2002 Feb;102(2):212-25. doi: 10.1016/s0002-8223(02)90050-7. PMID 11846115
- [Background] Subar AF, Thompson FE, Kipnis V, Midthune D, Hurwitz P, McNutt S, McIntosh A, Rosenfeld S. Comparative validation of the Block, Willett, and National Cancer Institute food frequency questionnaires : the Eating at America's Table Study. Am J Epidemiol. 2001 Dec 15;154(12):1089-99. doi: 10.1093/aje/154.12.1089. PMID 11744511
- [Background] Subar AF, Kipnis V, Troiano RP, Midthune D, Schoeller DA, Bingham S, Sharbaugh CO, Trabulsi J, Runswick S, Ballard-Barbash R, Sunshine J, Schatzkin A. Using intake biomarkers to evaluate the extent of dietary misreporting in a large sample of adults: the OPEN study. Am J Epidemiol. 2003 Jul 1;158(1):1-13. doi: 10.1093/aje/kwg092. PMID 12835280